CLINICAL TRIAL: NCT03777917
Title: Pilot Study to Assess the Effectiveness and Safety of Belotero Balance® Injection for Volume Augmentation of the Infraorbital Hollow
Brief Title: A Pilot Study to Assess the Effectiveness and Safety of Belotero Balance® Injection for Volume Augmentation of the Infraorbital Hollow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M930121001
Record Dates: First submitted 2018-12-04; First posted 2018-12-17 (Actual); Results first posted 2022-09-02 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Correction of Volume Loss in the Infraorbital Hollow Area

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Belotero Balance® (Experimental)
  Interventions: Device: Belotero Balance®
- No treatment (No Intervention)

INTERVENTIONS:
Device: Belotero Balance® — Belotero® Balance for infraorbital hollows. Mode of application: subdermal injection.
  Arms: Belotero Balance®

SUMMARY:
The pilot study aims to define safety, effectiveness, and patient-reported outcomes for Belotero Balance® use in the infraorbital hollows.

ELIGIBILITY:
Inclusion Criteria:

* Has right and left infraorbital hollow (IOH) volume deficit with a rating of 2 or 3 (moderate or severe) on the MIHAS.
* Has the same MIHAS score on both IOHs (i.e., IOHs are symmetrical).
* Is at least 22 years of age.

Exclusion Criteria:

* Ever been treated with fat injections or permanent and/or semi-permanent dermal fillers in the midfacial region.
* Received lower eyelid and/or malar region treatments with any absorbable or temporary fillers such as porcine-based collagen fillers, hyaluronic acid (HA) products, RADIESSE®, poly L-lactic acid (PLLA) or received mesotherapy treatment to the area within the past 24 months or plans to receive such treatments during participation in the study.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-12-27 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2020-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (3):
- United States (3):
  - Center for Sight, Merz Investigational Site #0010414, Sarasota, Florida
  - Private Practice, Merz Investigational Site #0010413, New York, New York
  - Center for Laser and Facial Surgery, Merz Investigational Site #0010353, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biesman B, Verma A, Cheng N, Duncan A. Development and Validation of a Photonumeric Scale for Evaluation of Infraorbital Hollowing. J Drugs Dermatol. 2023 Jan 1;22(1):74-81. doi: 10.36849/JDD.7191. PMID 36607759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 investigational sites in the United States.
Pre-assignment Details: A total of 66 participants were randomized.
Groups:
- Treatment With Belotero Balance®: IOH injected with Belotero Balance®.
- Untreated Control Group: No treatment.
Period: Overall Study
Arm/Group | Treatment With Belotero Balance® | Untreated Control Group
Started | 43 | 23
Safety Population (1 participant randomized into treatment group did not receive any treatment and was excluded from the safety population, and 1 participant randomized into the untreated group received Belotero Balance®.) | 43 | 22
Completed | 34 | 21
Not Completed | 9 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Lost to Follow-up | 6 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety population (SP) consisted of all randomized participants who received at least one study treatment in the active treatment group or who were randomized into the control arm.
Groups:
- Treatment With Belotero Balance®: Belotero Balance®, subcutaneous injection for IOHs.
- Total: Total of all reporting groups
Arm/Group | Treatment With Belotero Balance® | Untreated Control Group | Total
Number analyzed (Participants) | 43 | 22 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (12.6) | 47.3 (11.6) | 46.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 18 | 55
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 38 | 20 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 4 | 7
  White | 38 | 17 | 55
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Responder Rate Compared to the Untreated Control Group According to the Merz Infraorbital Hollow Assessment Scale (MIHAS).
Description: MIHAS was a 5 point scale ranging as: Grade 0 (none to minimal), Grade 1 (mild), Grade 2 (moderate), Grade 3 (severe), Grade 4 (extreme). Responder rate was defined as percentage of participants with treatment response who achieved greater than or equal to (>=) 1 grade improvement on both IOHs on the MIHAS.
Time Frame: Baseline up to Month 2
Population: The intent-to-treat (ITT) population consisted of all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment With Belotero Balance® | Untreated Control Group
Number analyzed (Participants) | 38 | 21
percentage of participants | 81.6 | 9.5
Statistical Analysis 1: Comparison: Treatment With Belotero Balance® vs Untreated Control Group; Test type: Superiority; p < 0.0001, Fisher Exact; The Fisher's exact test was used to test for the superiority of treatment (Belotero Balance®) over control; Difference in Response Rates = 72.1, 95% CI 2-sided [47.5 to 83.5] — Two-sided Newcombe confidence interval (CI) for the difference in response rates

2. Secondary Outcome: Change From Baseline in Rasch-Transformed Score for the Face-Q Satisfaction With Eyes
Description: The FACE-Q is a set of standardized patient-reported outcome scales for participants undergoing facial cosmetic procedures. The participants answered 7 questions of the FACE-Q satisfaction with eyes scale using a 4 point scale where: 1 (very dissatisfied), 2 (somewhat dissatisfied), 3 (somewhat satisfied), 4 (very satisfied). The sum scores of the FACE-Q satisfaction with eyes questionnaire and the Rasch-transformed scores ranging from 0 to 100 were summarized by treatment arm. Higher scores reflected a better outcome.
Time Frame: Baseline and Month 2
Population: The ITT population consisted of all randomized participants. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Treatment With Belotero Balance® | Untreated Control Group
Number analyzed (Participants) | 38 | 21
score on a scale | 28.8 [21.2 to 36.5] | 2.1 [-3.9 to 8.1]

3. Secondary Outcome: Global Aesthetic Improvement Scale (GAIS) Scores
Description: 7 point rating scale ranging from: +3 (very much improved), +2 (much improved), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), -3 (very much worse).
Time Frame: Baseline up to Month 2
Population: The ITT population consisted of all randomized participants. Here "overall number of participants analyzed" were participants who were evaluable for this outcome measure. As planned, this OM was evaluated only for participants treated with Belotero Balance®.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Belotero Balance®
Number analyzed (Participants) | 38
Participants
  Very Much Improved (+3) | 23
  Much Improved (+2) | 4
  Improved (+1) | 11
  No Change (0) | 0
  Worse (-1) | 0
  Much Worse (-2) | 0
  Very Much Worse (-3) | 0

4. Secondary Outcome: GAIS Scores as Assessed by Participants
Description: Participants evaluated their IOHs on 7 point rating scale ranging from: +3 (very much improved), +2 (much improved), +1 (improved), 0 (no change), -1 (worse), -2 (much worse), -3 (very much worse).
Time Frame: Baseline up to Month 2
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Belotero Balance®
Number analyzed (Participants) | 38
Participants
  Very Much Improved (+3) | 11
  Much Improved (+2) | 9
  Improved (+1) | 15
  No Change (0) | 2
  Worse (-1) | 1
  Much Worse (-2) | 0
  Very Much Worse (-3) | 0

5. Secondary Outcome: Responder Rate in the Treatment Group and the Untreated Control Group According to MIHAS as Assessed by Independent Panel Reviewers
Description: MIHAS was a 5 point scale ranging as: 0 (none to minimal), 1 (mild), 2 (moderate), 3 (severe), 4 (extreme). Responder rate was defined as percentage of participants with treatment response who achieved >=1 improvement on both IOHs compared to baseline. A participant was considered a responder if a treatment response of at least a 1-point change on both IOHs was determined by independent panel reviewers.
Time Frame: Baseline up to Month 2
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Treatment With Belotero Balance® | Untreated Control Group
Number analyzed (Participants) | 38 | 21
percentage of participants | 36.8 | 9.5

6. Secondary Outcome: Number of Participants Reporting One or More Device and/or Injection Related Treatment-emergent Adverse Events (TEAEs) and Device and/or Injection Related Serious TEAEs
Time Frame: Treatment Group: Baseline up to Month 13; Untreated Control Group: Baseline up to Month 2
Population: The SP consisted of all randomized participants who received at least one study treatment in the active treatment group or who were randomized into the control arm.
Measure: Count of Participants; unit: Participants
Groups:
- Treatment With Belotero Balance®: Belotero Balance®, subcutaneous injection at baseline for IOHs.
Arm/Group | Treatment With Belotero Balance® | Untreated Control Group
Number analyzed (Participants) | 43 | 22
Participants
  TEAEs | 2 | 0
  Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment Group : Baseline up to Month 13; Untreated Control Group: Baseline up to Month 2
Description: The investigator reported AEs systematically at each visit.
Arm/Group | Treatment With Belotero Balance® | Untreated Control Group
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/22
Serious Adverse Events (participants affected / at risk) | 1/43 | 0/22
Other Adverse Events (participants affected / at risk) | 0/43 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment With Belotero Balance® (N=43) | Untreated Control Group (N=22)
Retinal detachment (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03777917/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT03777917/SAP_001.pdf